CLINICAL TRIAL: NCT00053651
Title: Depression Intervention for Poor Pregnant Women
Brief Title: Prevention of Postpartum Depression in Low-Income Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21MH061555 (NIH); R21MH061555 (NIH); DSIR AT-AS
Record Dates: First submitted 2003-02-04; First posted 2003-02-05 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Survival Skills for Moms with New Babies

SUMMARY:
This study will determine whether a prevention program reduces the incidence of postpartum depression in pregnant women who receive public assistance and are at risk for postpartum depression.

DETAILED DESCRIPTION:
The impact of major depression in the postpartum period is profound, with considerable emotional pain for the new mother as well as disturbances in infant development. Unfortunately, few preventive interventions have been developed or systematically tested to reduce the risk of postpartum depression. An area of even greater neglect is the development of such an intervention for financially disadvantaged women who are at high risk for postpartum depression and for the disturbances associated with postpartum depression. This study will develop a psychosocial intervention for financially disadvantaged pregnant women at risk for postpartum depression.

Participants are randomly assigned to receive either the "Life at Home with a New Baby" intervention or care as usual. Women who receive the intervention join a counseling group in which information about mother-baby relationships is shared. This information is reinforced with a follow-up "booster" session after the infant is born. Participants are assessed at baseline, after the booster session (for the intervention condition) or after 2 weeks postdelivery (for the care as usual condition), and at 3 months postpartum. Depression levels and social adjustment are measured at baseline and 2 weeks after delivery. Functional status is also measured. A self-report questionnaire is completed by the mothers to measure parental distress, parent/child dysfunctional behavior, and difficult child interactions. At 3 months postpartum, a brief standardized interview is used to assess the presence of a depressive disorder.

ELIGIBILITY:
Inclusion criteria:

* Receive public assistance
* At risk for postpartum depression
* Pregnant women between 23-32 weeks gestation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250
Dates: Start 2001-09

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States